CLINICAL TRIAL: NCT00348166
Title: Does Undercorrection of Myopia Retard Myopia Progression Among Kindergarten
Brief Title: Does Undercorrection of Myopia Retard Myopia Progression Among Kindergarten Children?
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Stringent eligibility criterion caused difficulties in recruiting patients.
Sponsor: KK Women's and Children's Hospital (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: RAU/085/2005
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Refractive Error - Myopia
MeSH Terms: interventions — Cyclopentolate

INTERVENTIONS:
Drug: cyclopentolate

SUMMARY:
The purpose of this study is to find out if undercorrection of myopia slow down the progression of myopia in kindergarten children.

ELIGIBILITY:
Inclusion Criteria:

1. Children of chinese descent aged 5 - 6yrs
2. Refractive error of -1.00 to -3.00Ds
3. Less than 1.50 astigmatism in each eye. (No oblique axis)
4. Visual acuity is 6/6 or better in both eyes.
5. No binocular problems, no anisometropia >1.50D
6. Will be staying in S'pore for at least 2 years.

Exclusion Criteria:

-

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quah Boon Long, Principal Investigator — Singapore National Eye Centre